CLINICAL TRIAL: NCT05974839
Title: Effect of Ocrelizumab on Cortical Lesion Accumulation in Patients With Primary-progressive Multiple Sclerosis Participating in the ORATORIO: a Post-hoc Analysis of a Double-blind, Randomized, Phase 3, Placebo-controlled Study
Brief Title: Effect of Ocrelizumab on Cortical Lesion Accumulation in Patients With PPMS (ORATORIO-Cortical)
Acronym: ORATORIO-Cort
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 00007536
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ocrelizumab — Non-interventional

SUMMARY:
The goal of this non-interventional, observational study is to determine whether cortical pathology can be slowed down by use of ocrelizumab.

DETAILED DESCRIPTION:
To study the effect of ocrelizumab on cortical lesion accumulation in patients with primary-progressive multiple sclerosis participating in the ORATORIO: a post-hoc analysis of a double-blind, randomized, phase 3, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Patient participating in the ORATORIO study
* MRI scans available at baseline
* Presence of T2-weighted image (WI) (FLAIR, T2/PD), and 2D/3D T1-WI at baseline

Exclusion Criteria:

- None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Primary Progressive Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Cortical lesion number accumulation | 5 years
  Cortical lesion accumulation as measured using MRI between subjects on placebo and subjects who took ocrelizumab.

SECONDARY OUTCOMES:
Cortical lesion number accumulation and disability. | 5 years
  Cortical lesion number accumulation as measured by MRI for subjects who developed disability over the course of the placebo-controlled phase of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No